CLINICAL TRIAL: NCT06843837
Title: The Effect of Sweet Orange Aromatherapy on Anxiety and Pulse Level of Nurse Students During IV Cannula Placement Skill Process
Brief Title: The Effect of Sweet Orange Aromatherapy on Anxiety and Pulse Level of Nurse Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, seher ÇEVİK, Assistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: inonu university 2
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: University Students
Keywords: Sweet orange aromatherapy; Nursing students; IV cannulation skill; Anxiety; Heart rate
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental model
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In this study, sweet orange essential oil was applied to reduce anxiety levels and physiological responses of nursing students during IV cannulation skill practice. The study data were collected in the intravenous (IV) access rooms of Fırat University Medical Center Hospital's outpatient clinic. There are two IV access rooms on the outpatient clinic floor, one of which was randomly assigned to the control group and the other to the experimental group. After administering pre-tests (Participant Information Form, Pulse Monitoring Form, and State-Trait Anxiety Inventory [STAI]), students were instructed to perform IV cannulation on the assigned patient. A cotton ball infused with three drops of sweet orange essential oil was held 4 to 5 cm away from the student's nose, and they were instructed to breathe slowly for five minutes. After this, the students were asked to perform IV cannulation on the patient.
  Interventions: Other: Sweet orange essential oil aromatherapy
- control (No Intervention)

INTERVENTIONS:
Other: Sweet orange essential oil aromatherapy — The sweet orange essential oil used in the study was prepared by the Food Engineering Department of Fırat University. To obtain the essential oil used for aromatherapy in this study, the peels of Citrus sinensis sweet oranges were utilized. The orange peels were cut into small pieces of approximately 3-5 mm in size, placed into a boiling flask, and distilled water was added. Based on the analysis results, the percentage composition of the total essential oil fatty acids was determined. The chemical composition analysis revealed that D-limonene was the major component, comprising 90% of the total oil. The oil is 100% pure essential oil, containing up to 90% D-limonene, along with citral and linalool. A cotton ball infused with three drops of sweet orange essential oil was held 4 to 5 cm away from the student's nose, and they were instructed to breathe slowly for five minutes. After this, the students were asked to perform IV cannulation on the patient.
  Other Names: Sweet orange aromatherapy
  Arms: Intervention

SUMMARY:
This randomized controlled study examined the effect of sweet orange essential oil aromatherapy on reducing anxiety experienced by nursing students during the IV cannulation process. First-year nursing students from a university in eastern Turkey participated in the study. According to the sample size determined by G*Power analysis, 100 students were randomized, and the study was completed with 47 students in the experimental group and 48 students in the control group.

All students were taught IV cannulation skills theoretically and practically. Subsequently, students in the experimental group performed IV cannulation on real patients after receiving aromatherapy. Data were collected using a Personal Information Form, a Pulse Monitoring Form, and the State-Trait Anxiety Inventory (STAI).

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the effectiveness of sweet orange essential oil aromatherapy in reducing anxiety among nursing students during the IV cannulation procedure. The study was conducted with first-year nursing students enrolled in the nursing department of a university in eastern Turkey. The sample size was determined using G*Power analysis, and a total of 100 students were randomized into two groups. The study was completed with 47 students in the experimental group and 48 students in the control group.

All participants received standardized theoretical and practical training on IV cannulation. Following the training, students in the experimental group were exposed to sweet orange essential oil aromatherapy before performing IV cannulation on real patients, while those in the control group proceeded with the procedure without aromatherapy intervention.

Data collection tools included a Personal Information Form, a Pulse Monitoring Form to track physiological responses, and the State-Trait Anxiety Inventory (STAI) to assess anxiety levels. The study aimed to determine whether aromatherapy could serve as an effective non-pharmacological strategy for alleviating procedural anxiety among nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being actively enrolled in school, not having performed an IV cannulation before, taking the Basic Principles and Fundamentals in Nursing I course, and not having any health issues that would prevent inhaling sweet orange oil.

Exclusion Criteria:

* Not volunteering to participate in the study, not being actively enrolled in school, and having any health issues that would prevent inhaling sweet orange oil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) | 3 month
  developed by Spielberger and colleagues in 1970, was adapted into Turkish by Öner and LeCompte. This four-point Likert scale consists of 20 short statements, 10 of which are reverse-coded. In the scale, the total score from the straightforward statements is subtracted from the total score of the reverse-coded statements, and a fixed number, 50, is added to the result. The scores obtained through this method range from 20 to 80, with scores between 20-39 indicating low, 40-59 indicating moderate, and 60-79 indicating high levels of anxiety. An increase in the score indicates a rise in the individual's anxiety level. The reliability coefficients of the scale range from 0.94 to 0.96 (Spielberger et al., 1970; Öner and LeCompte, 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' data were collected for research purposes only according to the ethical principle of confidentiality and protection. Therefore, it cannot be shared.